CLINICAL TRIAL: NCT01359475
Title: Phase 3- Clinical Trial on Children. PROTOCOL 465-549
Brief Title: A Clinical Trial of an Acetal Resin Crown for Restoration of Primary Molars
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Uri Zilberman (Other)
Collaborators: Uri Zilberman (Unknown)
Responsible Party: Sponsor-Investigator, Uri Zilberman, Head of Dentistry Unit, Barzilai Medical Center
Organization: Barzilai Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMC1505CTIL; PROTOCOL 465-549 (Other: LD Caulk, Usa)
Record Dates: First submitted 2011-05-15; First posted 2011-05-24 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Other Unsatisfactory Restoration of Tooth
Keywords: Acetal crowns; Primary molars; The retention of acetal crowns in primary dentition; Color changes of acetal crowns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acetal crown (Experimental): Clinical performance of acetal crowns for treatment of primary molars
  Interventions: Procedure: Acetal crown, LD Caulk ltd, USA

INTERVENTIONS:
Procedure: Acetal crown, LD Caulk ltd, USA — Experimental trial of preformed acetal crowns for primary molars
  Other Names: Prefabricated crowns for primary molars

SUMMARY:
Preformed stainless steel crowns have been used in Pediatric Dentistry to restore badly broken down primary teeth since 1950. They are generally considered more expedient to place than large multi-surface amalgam or composite restorations and have a longer life. They have been used successfully in clinical practice for many years and have presented little in the way of adverse events. The major drawback is the poor esthetics along with lingering concerns over potential health hazards associated with the nickel content. Several attempts have been made to improve upon the esthetics of stainless steel crowns such as veneering the buccal and occlusal surfaces and substituting composite resin for the entire crown, but to date none of these approaches have been very successful.

Acetal resin has been used in a number of applications in medicine and dentistry, and recently has met with early success when tested as a substitute for stainless steel crowns. It has a number of excellent physical and mechanical properties including a low coefficient of friction, good wear resistance, high fatigue resistance, good impact strength and resistance to creep.

The purpose of this trial is to compare the clinical performance of preformed acetal resin crowns and preformed stainless steel crowns.

2.0 OBJECTIVES

The objective of this study is to compare the clinical performance of acetal resin crowns with preformed stainless steel crowns when used to restore primary molar teeth.

DETAILED DESCRIPTION:
STUDY POPULATION

A minimum of 25 subjects contributing a minimum of 40 acetal crowns ( on primary molar teeth will be recruited from the patient pool of the pediatric dentistry clinic at Barzilai Medical Center, Ashkelon and enrolled into the study. A maximum of four crowns will be placed in any subject. It is estimated that it will take approximately 14 weeks to place all crowns and complete the baseline examination.

ELIGIBILITY:
Inclusion Criteria:

* Patients of record at the pediatric dentistry clinic at Barzilai Medical Center, Ashkelon
* Ages 3-8 (inclusive)
* In need of at least one Stainless Steel Crown on either a first or second primary molar

Exclusion Criteria:

* Medically compromising condition
* Informed consent not given
* Teeth with proximal space closures of sufficient magnitude to preclude placement of a test crown

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Retention of acetal crowns for primary molars | two years
  Number of patients with adverse events

SECONDARY OUTCOMES:
Color stability of acetal crown | two years
  Change from baseline color of acetal crowns

CONTACTS AND LOCATIONS:
Overall Officials: Uri L Zilberman, DMD, PhD, Principal Investigator — Barzilai Medical Center
Locations (1):
- Pediatric Dental Clinic, BarzilaiMC, Ashkelon, Israel